CLINICAL TRIAL: NCT03678506
Title: APIDULCIS: Extended Anticoagulation With Low-dose Apixaban After a Standard Course Anticoagulation in Patients With a First Venous Thromboembolism Who Have Positive D-dimer
Brief Title: Apixaban for Extended Anticoagulation (APIDULCIS)
Acronym: APIDULCIS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was interrupted after a planned interim analysis for the high rate of primary outcomes (7.3%; 95% confidence interval [CI], 4.5-11.2)
Sponsor: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAA I1. 7-2017 (APIDULCIS); 2017 002340 32 (EudraCT Number)
Record Dates: First submitted 2018-09-08; First posted 2018-09-19 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Venous Thromboembolism; Anticoagulants
Keywords: Venous thromboembolism; D-Dimer; Apixaban; Extended treatment
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: The patients included in the study will receive a serial determination of D-dimer assay (a maximum of four determinations in case of negative results).The D-dimer measurements should be performed at the moment of patient screening, when patients still assume their anticoagulant treatment (T0), at 15±2 days (T1), 30±4 days (T2), and 60±5 (T3) days after their anticoagulant treatment has been stopped. At the first positive D-dimer result patients resume anticoagulation with apixaban 2.5 mg bis in die for the next 18 months. Patients with negative D-Dimer results at all determinations stop anticoagulation definitely and will followed up for the next 18 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive D-Dimer (Experimental): At the first positive D-dimer results (during anticoagulation or after its temporary withdrawal) the patients are invited to assume Eliquis (apixaban) 2.5 mg twice daily, and continue this therapy for the following 18 months.
  Interventions: Drug: Apixaban
- Negative D-Dimer (No Intervention): Patients with persistently negative results at the four serial D-dimer measurements, stay definitively without anticoagulation and discouraged to resume any antithrombotic drug for secondary VTE prevention.

INTERVENTIONS:
Drug: Apixaban — Apixaban 2.5 mg x 2 will be administered to patients with positive D-dimer results
  Other Names: Apixaban and positive d-dimer
  Arms: Positive D-Dimer

SUMMARY:
The study aims at optimizing the long-term and extended management of patients with a first episode of venous thromboembolism (proximal deep vein thrombosis with or without pulmonary embolism) (VTE). Patients at high risk of recurrence (with altered D-dimer test), who had received anticoagulation (whatever the drug used) for 12-15 months after the first episode of thrombosis, will be treated with Apixaban 2,5 mg x 2 for 18 months as extended treatment. Patients at low risk, with normal D-dimer test, will stop anticoagulation definitely.

DETAILED DESCRIPTION:
This prospective cohort study aims to assess the efficacy and safety of a management procedure to decide on giving or not an extended anticoagulation (administering apixaban 2 2.5 mg twice daily ) to outpatients with a single episode of proximal deep vein thrombosis of the lower limbs and/or pulmonary embolism who had received 12-15 months of anticoagulation (whatever the anticoagulant drug used). The study seeks to assess whether a management procedure involving D-dimer testing assessment can identify a subset of subjects at low risk of recurrence in whom an extended anticoagulation can be safely avoided.

ELIGIBILITY:
Inclusion Criteria:

* First unprovoked Venous Thromboembolic Event
* Venous Thromboembolic events associated with one or more risk factors that are no longer present
* Age older than 18 or younger than 75 years
* Capacity to give written informed consent

Exclusion Criteria:

* A) Exclusion criteria regarding the index event
* Events usually associated with low risk of recurrence
* Deep vein thrombosis/ Pulmonary embolism occurred within 3 months from major surgery or major trauma
* Isolated Distal deep vein thrombosis (thrombosis of calf veins)
* Events associated with a very high risk of recurrence or occurrence of life-threatening recurrent events

  * Pulmonary Embolism episode with shock or life-threatening
  * Isolated pulmonary embolism with a systolic pulmonary artery pressure > 60 mmHg at presentation
  * Deep vein thrombosis/ Pulmonary embolism associated with active cancer, antiphospholipid syndrome or long-standing medical illnesses
  * More than one idiopathic event
* Index venous thromboembolic event in different sites than deep veins of the lower limbs or pulmonary arteries

B) Exclusion criteria present at the moment of patients' screening:

* Age younger than 18 or older than 75 years
* More documented unprovoked venous thromboembolic episodes
* Pregnancy or puerperium
* Severe post-thrombotic syndrome (≥ 15 points at the Villalta score)
* Solid neoplasia or blood disease in active phase or requiring chemotherapy/radiotherapy
* All the clinical conditions requiring prolonged treatment with Low Molecular Weight Heparin
* Presence of overt, active chronic diseases (i.e. inflammatory bowel disease)
* Known serious thrombophilic alterations:

  * deficiencies of natural anticoagulants (Antithrombin, Protein C, Protein S)
  * homozygosity for Factor V Leiden or Factor II G20210A mutations
  * double heterozygosity
* Presence of antiphospholipid syndrome
* Presence of vein cava filter
* Concomitant conditions (such as atrial fibrillation) requiring indefinite anticoagulation
* Severe cardio-respiratory insufficiency (NYHA 3 or 4)
* Any absolute contraindications to anticoagulation treatment
* Any other contraindications to Apixaban as per local SmPC
* Life expectancy shorter than 1 year
* Refuse interruption of anticoagulation to perform serial D-dimer assessment
* Geographically inaccessible location
* Inability or refusal to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number and rate of patients with confirmed recurrent VTE and VTE-related death (efficacy). | From date of enrollment until the date of first documented event assessed up to 18 months
  The occurrence of proximal deep vein thrombosis with or without pulmonary embolism (new or recurrent episode) wil be recorded in all patients
Number and rate of major Bleeding events (defined according to International Society on Thrombosis and Haemostasis guidelines (safety) | From date of enrollment until the date of first documented event assessed up to18 months
  Fatal bleeding; intracranial; intraspinal; intraocular; pericardial; intra-articular; intramuscular with compartment syndrome; retroperitoneal,; acute clinically overt bleeding will be recorded in all patients

SECONDARY OUTCOMES:
Number of and rate of thromboembolic events | From date of enrollment until the date of first documented event assessed up to 18 months
  Transient ischemic attack (TIA), Stroke, Myocardial infarction will be recorded in all patients
Presence of severe post-thrombotic syndrome according to Villalta Score | 18 months
  Patient with deep vein thrombosis as index event will be evaluated, at the and of follow-up, applying Villalta score, commonly used to diagnose post-thrombotic syndrome in the subacute phase of thrombosis. The presence of venous ulcer of the leg or a score > of 15 points indicate the occurrence of severe post-thrombotic syndrome. The maximum score is 33. The score from 5 to 9 points indicate mild post-thrombotic syndrome and from 10 to 15 points indicate moderate post-thrombotic syndrome
Number and rate of non major bleeding complications | From date of enrollment until the date of first documented event assessed up to18 months
  In all patients will be recorded any sign or symptom of hemorrhage that does not fit the criteria for the definition of major bleeding but does meet at least one of the following criteria: 1)requiring medical intervention by a healthcare professional; 2) leading to hospitalization or increased level of care;3) prompting a face to face evaluation
Number and rate of dead patients (overall mortality) | From date of enrollment until the date of first documented event assessed up to 18 months
  VTE-related death; cardiovascular related-death; bleeding-related death; death for: cancer, infectious disease and unknown cause; sudden death will be recorded in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Poli, MD, Study Director — Azienda Ospedaliero-Universitaria Careggi, Firenze, Italy
Locations (1):
- Daniela Poli, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after the publication of global results of the study or after 18 months from the enrollment of the last patients
Access Criteria: Data access requests will be reviewed by the Scientific board of the study.

REFERENCES:
- [Derived] Palareti G, Poli D, Ageno W, Legnani C, Antonucci E, Bucherini E, Testa S, Paoletti O, Chistolini A, Serrao A, Martinelli I, Bucciarelli P, Falanga A, Tosetto A, Sarti L, Mastroiacovo D, Cosmi B, Visona A, Santoro RC, Zanatta N, Grandone E, Bertu L, Pengo V, Caiano L, Prandoni P. D-dimer and reduced-dose apixaban for extended treatment after unprovoked venous thromboembolism: the Apidulcis study. Blood Adv. 2022 Dec 13;6(23):6005-6015. doi: 10.1182/bloodadvances.2022007973. PMID 35914222

DOCUMENTS (2):
  • Study Protocol (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03678506/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03678506/SAP_001.pdf